CLINICAL TRIAL: NCT05250414
Title: Cochlear Implantation in the Single-Sided Deafness in the Medicare Population
Brief Title: Single-Sided Deafness in the Medicare Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-EL SSD CMS
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Procedure (Other)
  Interventions: Device: MED-EL Cochlear Implant System

INTERVENTIONS:
Device: MED-EL Cochlear Implant System — Cochlear implant and audio processor

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of cochlear implantation in adults 65 years of age and older.

DETAILED DESCRIPTION:
The study will be conducted as a single-subject, repeated measures, multi center study at 3 sites. Fifteen subjects will be enrolled in this study. Three centers in the United States and Canada will recruit subjects into this study. Study subjects will be followed for 12 months post-implantation of the device.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older at the time of implantation
* Unilateral profound hearing loss, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 90 dB or greater in the ear to be implanted
* Sensorineural hearing loss in the ear to be implanted, as defined by an air-bone gap less than or equal to 10 dB at two or more frequencies out of 500, 1000, 2000, and 4000 Hz
* Normal or near-normal hearing in the non-implanted ear, as defined by a pure-tone average (500, 1000, 2000, and 4000 Hz) of 30 dB or less
* Word recognition in the ear to be implanted of 5% or less on CNC word score in quiet
* Previous experience with an appropriately-fit CROS, BI-CROS, bone conduction, or traditional hearing aid, as deemed appropriate by investigator
* Fluent in English

Exclusion Criteria:

* Duration of profound hearing loss of 10 years or more
* Sudden onset of hearing loss within six months of implantation
* Evidence of non-functional cochlear nerve or other retrocochlear hearing loss
* Evidence of severe cochlear malformation (i.e., common cavity or ossification)
* External or middle ear infection
* Suspected cognitive concern
* Other medical contraindication for surgery or anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Performance of the Cochlear Implant System will be assessed through speech perception testing in noise completed through one year (12 months) post implantation. | One year (12 months) post implantation
  The primary effectiveness endpoint will be change on speech in noise when speech is presented to the front and noise is presented to the acoustic hearing (contralateral) ear. The pre-operative, best aided score will be compared to the 6-month and 12-month CI score for AzBio sentences in noise (range of score 0-100, higher score is better). Improvement is defined as greater than or equal to 10 percentage points.

SECONDARY OUTCOMES:
Performance of the Cochlear Implant System will be summarized through speech perception testing in noise completed through one year (12 months) post implantation. | One year (12 months) post implantation
  Speech in noise in two spatial conditions will demonstrate similar performance from the pre-operative, best-aided score to the CI score at 6- and 12-months post activation. AzBio sentence in noise score will be summarized for two conditions: speech and noise presented from the front as well as speech presented to the front and noise presented to the CI ear. (Range of score 0-100, higher score is better)
Performance of the Cochlear Implant System will be assessed through speech perception testing in quiet completed through one year (12 months ) post implantation. | One year (12 months) post implantation
  Speech perception in quiet will be summarized for the CI ear as well as the contralateral ear at the pre-operative, 6-month, and 12-month intervals. The CI ear is expected to demonstrate improvement (greater than or equal to 10 percentage point change), while the contralateral ear is expected to demonstrate no change. (Range of score 0-100, higher score is better)
Subjective benefit of the Cochlear Implant System will be assessed through one year (12 months) post implantation. | One year (12 months) post implantation
  Subjective data will be collected via the Speech, Spatial, and Qualities of Hearing Scale (SSQ). Responses will be summarized from the pre-operative, 6-month, and 12-month intervals. (Range of score 0-10, lower score is better)
Safety will be evaluated for all study subjects through one year (12 months) post implantation. | One year (12 months) post implantation
  Safety will be assessed by collecting and reporting device-related adverse events occurring throughout the study. This will be summarized and reported as the number and proportion of subjects experiencing an adverse device event.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of North Carolina, Chapel Hill, North Carolina
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Arndt S, Laszig R, Aschendorff A, Hassepass F, Beck R, Wesarg T. Cochlear implant treatment of patients with single-sided deafness or asymmetric hearing loss. HNO. 2017 Aug;65(Suppl 2):98-108. doi: 10.1007/s00106-016-0297-5. PMID 28188428
- [Background] Buss E, Dillon MT, Rooth MA, King ER, Deres EJ, Buchman CA, Pillsbury HC, Brown KD. Effects of Cochlear Implantation on Binaural Hearing in Adults With Unilateral Hearing Loss. Trends Hear. 2018 Jan-Dec;22:2331216518771173. doi: 10.1177/2331216518771173. PMID 29732951
- [Background] Mertens G, De Bodt M, Van de Heyning P. Evaluation of Long-Term Cochlear Implant Use in Subjects With Acquired Unilateral Profound Hearing Loss: Focus on Binaural Auditory Outcomes. Ear Hear. 2017 Jan/Feb;38(1):117-125. doi: 10.1097/AUD.0000000000000359. PMID 27513880
- [Background] Niparko JK, Cox KM, Lustig LR. Comparison of the bone anchored hearing aid implantable hearing device with contralateral routing of offside signal amplification in the rehabilitation of unilateral deafness. Otol Neurotol. 2003 Jan;24(1):73-8. doi: 10.1097/00129492-200301000-00015. PMID 12544032
- [Background] Van de Heyning P, Vermeire K, Diebl M, Nopp P, Anderson I, De Ridder D. Incapacitating unilateral tinnitus in single-sided deafness treated by cochlear implantation. Ann Otol Rhinol Laryngol. 2008 Sep;117(9):645-52. doi: 10.1177/000348940811700903. PMID 18834065
- [Background] Vermeire K, Van de Heyning P. Binaural hearing after cochlear implantation in subjects with unilateral sensorineural deafness and tinnitus. Audiol Neurootol. 2009;14(3):163-71. doi: 10.1159/000171478. Epub 2008 Nov 13. PMID 19005250